CLINICAL TRIAL: NCT03866486
Title: Impact of IntraVascular UltraSound Guidance on the Outcomes of Xience Prime Stents in Long Lesions (IVUS-XPL Study): Retrospective and Prospective Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-1153
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Myocardial Ischemia(Implanted Drug-eluting Stents Because of Ischemic Heart Disease(Stable Angina, Acute Coronary Syndrome))
Keywords: Clinical outcome; IVUS; Stent
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVUS-guidance group: The patients who underwent drug-eluting stents implantation with IVUS guidance.
- Angiography-guidance group: The patients who underwent drug-eluting stents implantation with angiography guidance without IVUS.

SUMMARY:
The investigator aimed to evaluate the long-term (up to 10 years) follow-up of the patients who enrolled the IVUS-XPL study (Impact of IntraVascular UltraSound Guidance on the Outcomes of Xience Prime Stents in Long Lesions), which was shown the superiority of IVUS-guided stent implantation at 1 year in terms of major adverse cardiac events.

DETAILED DESCRIPTION:
The investigator will follow-up (up to 10 years) the patients who enrolled the IVUS-XPL study (Impact of IntraVascular UltraSound Guidance on the Outcomes of Xience Prime Stents in Long Lesions).

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients who enrolled in the XPL-IVUS study.
* 2. Provision of informed consent

Exclusion Criteria:

* 1. This observational study does not have any specific exclusion criteria.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who enrolled in the previous IVUS-XPL study. In the IVUS-XPL trial, the patients who implatned drug-eluting stents because of ischemic heart disease (stable angina, acute coronay syndrome) were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The composite of major adverse cardiac events, including cardiac death, target lesion-related myocardial infarction, or ischemia-driven target lesion revascularization at 5 years and at 10 years | At 5 years
  Major adverse cardiac events will be included the composite of cardiac death, target lesion-related myocardial infarction, or ischemia-driven target lesion revascularization.
The composite of major adverse cardiac events, including cardiac death, target lesion-related myocardial infarction, or ischemia-driven target lesion revascularization at 5 years and at 10 years | At 10 years
  Major adverse cardiac events will be included the composite of cardiac death, target lesion-related myocardial infarction, or ischemia-driven target lesion revascularization.

SECONDARY OUTCOMES:
Cardiac death at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Cardiac death at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
All-cause of death at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
All-cause of death at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Target-lesion related myocardial infarction at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Target-lesion related myocardial infarction at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Any myocardial infarction at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Any myocardial infarction at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Target-lesion revascularization at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Target-lesion revascularization at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Any revascularization at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Any revascularization at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Target-lesion related stent thrombosis at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Target-lesion related stent thrombosis at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Any stent thrombosis at 5 years | At 5 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.
Any stent thrombosis at 10 years | At 10 years
  Secondary outcome will include both the each component of primary outcome and non-target lesion-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Myeong-Ki Hong, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Hong SJ, Mintz GS, Ahn CM, Kim JS, Kim BK, Ko YG, Kang TS, Kang WC, Kim YH, Hur SH, Hong BK, Choi D, Kwon H, Jang Y, Hong MK; IVUS-XPL Investigators. Effect of Intravascular Ultrasound-Guided Drug-Eluting Stent Implantation: 5-Year Follow-Up of the IVUS-XPL Randomized Trial. JACC Cardiovasc Interv. 2020 Jan 13;13(1):62-71. doi: 10.1016/j.jcin.2019.09.033. PMID 31918944